CLINICAL TRIAL: NCT00889161
Title: Curcumin in Pediatric Inflammatory Bowel Disease: A Forced Dose Titration Study
Brief Title: Curcumin in Pediatric Inflammatory Bowel Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: David Suskind, MD, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Curcumin-1; 1UL1RR025014-01 (NIH)
Record Dates: First submitted 2009-04-24; First posted 2009-04-28 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Inflammatory Bowel Disease; Ulcerative Colitis; Crohn's Disease
Keywords: Crohn's disease; ulcerative colitis; curcumin; pediatric; inflammatory bowel disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease | interventions — Curcumin

INTERVENTIONS:
Drug: Curcumin — Initial dosage of 500mg twice a day for 3 weeks. Using the forced dose titration design, dose will be titrated up to 1g twice a day at Week 3 for a total of three weeks and then titrated again to 2g twice a day at Week 6 for three weeks.

SUMMARY:
This is a single center, open label forced dose titration study designed to determine the tolerability of curcumin in pediatric patients with inflammatory bowel disease (IBD). This study will provide initial tolerability and safety data in pediatric patients with IBD. Twenty patients with IBD in remission or with mild disease (score <34 on PUCAI or score <30 on the PCDAI) on sulfasalazine or mesalamine aged 8 to 18 years will be enrolled into this study. Each patient will participate in the study for nine weeks. From this study an appropriate dosage will be determined to proceed with a double blinded placebo controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents eight to eighteen years old
* Diagnosis of inflammatory bowel disease (IBD) made by a pediatric gastroenterologist based upon history, physical examination, laboratory/radiological studies and gastrointestinal histology
* Mild disease or in clinical remission based upon PUCAI or PCDAI score (score <34 on the PUCAI or score <30 on the PCDAI)
* Parent/guardian and participant must be able to attend study visits at screening, baseline, and weeks three, six, and nine
* Patient must be on a stable dose of IBD medications for at least 3 months
* Patient must be able to swallow study medication

Exclusion Criteria:

* Abnormal laboratory values as defined in the protocol
* History of increased gastrointestinal symptoms ("flare") in the last 3 months
* Current use (past use of these medications is not an exclusion) of medications such as azathioprine, methotrexate or 6-mercaptopurine used to treat IBD
* Current use (past use of these medications is not an exclusion) of medications or over-the-counter treatments including but not limited to aspirin, NSAID, botanical treatments (ginger, feverfew, yellow clover, Salix species, Populus species, Betula species, and Gaultheria species), essential fatty acids (flax oil and fish oil). Allowed supplementation includes multivitamin, vitamin D & calcium, folate and vitamin B12, and Iron.
* Other serious medical conditions such as neurological, liver, kidney, auto- immune or systemic disease.
* History of gastrointestinal surgery or planned gastrointestinal surgery in the future.
* Tobacco, alcohol, or illicit drug abuse
* Planned surgery during the potential study participation time
* Inability to swallow study medication

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine the tolerability of curcumin in pediatric patients with inflammatory bowel disease. | 9 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Suskind, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hosptial, Seattle, Washington, United States

REFERENCES:
- [Derived] Suskind DL, Wahbeh G, Burpee T, Cohen M, Christie D, Weber W. Tolerability of curcumin in pediatric inflammatory bowel disease: a forced-dose titration study. J Pediatr Gastroenterol Nutr. 2013 Mar;56(3):277-9. doi: 10.1097/MPG.0b013e318276977d. PMID 23059643